CLINICAL TRIAL: NCT00993122
Title: Phase 2 Randomized Multicenter Controlled Study of Ribavirin Pre-treatment (8 Weeks) Followed by Standard Therapy With Ribavirin and Pegylated Interferon (48 Weeks) in Transplanted Patients With Recurrence of Chronic Hepatitis C
Brief Title: Ribavirin Pre-treatment Followed by Combined Standard Therapy in Hepatitis C Virus (HCV) Recipients
Acronym: RBV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Manuela Merli, professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ribavirin Pre-treatment
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C
Keywords: pre treatment; therapy compliance; SVR; sustained virological response; TH1 TH2 ratio
MeSH Terms: conditions — Hepatitis C; Patient Compliance | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ribavirin pre-treatment (Active Comparator): patient will receive ribavirin in monotherapy for 8 weeks before the combined 48 weeks antiviral therapy
  Interventions: Drug: ribavirin pre-treatment
- combined stardard therapy (Active Comparator): patients will receive the standard combined therapy with ribavirin and pegylated interferon for 48 weeks
  Interventions: Drug: ribavirin pre-treatment

INTERVENTIONS:
Drug: ribavirin pre-treatment — patients receive ribavirin (10,4 mg/kg/day) and pegylated interferon alfa-2b (1,5 mcg/kg/week).Pre-treatment arm will receive a 8-week monotherapy treatment with only ribavirin (same dosage) and the controlled arm will receive 48 week of standard combined therapy (ribavirin plus pegylated interferon)
  Other Names: ribavirin pre treatment; ribavirin priming; Recurrence of hepatitis c; hepatitis c; transplanted patients; ribavirin; HCV

SUMMARY:
The results of antiviral therapy in patients with recurrent hepatitis C after liver transplantation are lower than standard. Ribavirin has immune-modulating effects and seems to be crucial to optimize viral treatment. The aim of this multicenter controlled study is to examine the effect of Ribavirin pre-treatment preceding the combination therapy with peginterferon plus ribavirin on the sustained virological response.

DETAILED DESCRIPTION:
Ribavirin Pre-Treatment Study Protocol

1. Introduction:

   * Recurrence of hepatitis C infection and liver transplant:

   Recurrence of hepatitis C after liver transplant is almost universal. After liver transplantation, the progression of chronic hepatitis C is more aggressive and an high percentage of recipients develop cirrhosis and rapid liver decompensation (1). Recent studies have shown that the long-term-survival-rate is significantly lower compared with non-HCV infected recipients (2). Other studies founded that antiviral treatment improves survival in these patients. Thus, the treatment of hepatitis C patients after LT is a priority for transplant units.

   To date, the rate of sustained virologic response (SVR) in patients with recurrent hepatitis C after liver transplantation is about 20% with standard IFN and increases to 30% with pegylated IFN and Ribavirin (3). Lack in tolerability and low compliance to the antiviral therapy may represent an important limiting factor in order to improve the SVR. Severe myelosuppression is frequent in these patients, due to the additional effect of immunosuppressive therapy, being an additional reason to reduce antiviral drug dosage (3).
   * Ribavirin:

   Recent studies have evaluated the effects of a ribavirin priming before the standard combined antiviral therapy in immuno-competent patients with chronic hepatitis C (4-7). The conclusion of these studies may suggest that ribavirin pre-treatment may be a way to improve the SVR.
2. Aim of the study:

   The study is a randomized un-blind multicenter project to compare the efficacy of antiviral treatment with a RBV priming vs standard antiviral treatment in patients with recurrent hepatitis C after liver transplantation.

   Ribavirin pre-treatment may:
   * Ameliorate therapy-compliance
   * Avoid a concomitant drugs-related hematological side effects
   * Modify the intra-hepatic cytokine pattern toward a better antiviral action
   * Improve the SVR.

   This controlled trial is not sponsored by a drug company.
3. Patients:

   The protocol of the study needs to be approved by the local ethic committee. Patients are enrolled in the study after been informed of the purpose and protocol of treatment and need to sign a written informed consent.
4. Statistical analysis, sample size and randomization:

   Sample size calculations were performed using EVR as the primary outcome measure. We assumed that 48 weeks intended treatment with pegylated interferon and ribavirin in transplant patients with recurrent hepatitis C induced EVR in about 60% of patients (10). In our pilot study ribavirin priming followed by 48 weeks of pegylated interferon and ribavirin obtained EVR in 92% of patients. To show an improvement of EVR from 60 to 92% , assuming an alpha level of 0.05, and 90% power ( beta =0.20) fifty patients per group are needed.

   Patients will be randomized after inclusion in the study, using an opaque envelope technique to be assigned to their treatment by a predetermined sequence at the Coordinator Center. Randomization will be stratified for genotype 1 and non1 to decrease the likelihood that uneven distribution of underlying disease severity would bias the results. Randomization will occur in blocks of four.
5. Definitions:

   The following definitions are going to be used; during the study:
   * Rapid Virological Response: complete viral clearance at week 4
   * Early Virologic Response: viral reduction > 2 log after 12 weeks of combined therapy.
   * Complete Early Virological Response: complete viral clearance after 12 weeks of combined therapy.
   * End of treatment Virologic Response: complete viral clearance at the end of the treatment period
   * Sustained Virologic Response: complete viral clearance 24 weeks after the end of treatment
   * Non Responder: Absence of virological response after 12 weeks
   * Relapse: recurrence of viral replication after a complete clearance during treatment time or after the conclusion of it.
6. Protocol of the study:

Basal Evaluation:

* Liver biopsy within the last 6 months
* Complete biochemical assessment (liver function tests, renal function, blood tests, levels of immunosuppressive therapy)
* HCV-RNA quantitative determination

Randomization: Patient are randomized to treatment A or Treatment B):

* Treatment A:

Pre-treatment:

Ribavirin is started at 600 mg/day (or 400mg/ day if < 60 kg) and increased to 10,4 mg/kg within week 2, the therapy is continued for 8 complete weeks.

Biochemical assessment is repeated at week 2, 4, 8. Samples are stored at the same times.

HCV-RNA quantitative determination is repeated at week 8. Drug reduction is allowed when hemoglobin level is below 10 g/dL though EPO administration or whenever it is considered necessary.

Combined antiviral therapy:

For 48 weeks patients are treated with Ribavirin (same dosage) and IFN alfa2b (1,5 mcg/kg/week).

Patients are followed monthly or more frequently if required. Biochemical and virological assessment is recorded at week 4, 12, 24, 48. Surveillance is performed for any collateral effects and dose adjustment or growth factor need.

Ribavirin reduction is required when hemoglobin level is below 10 g/dL though EPO use.

IFN weekly administration should be reduced when neutrophiles count is < 750 in spite of G-CSF administration.

IFN interruption is required when neutrophiles are < 500 or platelets are < 35000.

* Treatment B:

For 48 weeks patients are treated with Ribavirin (10 mg/kg ) and pegylated IFN alfa2b weekly.

Ribavirin is started at 600 mg/day and increased to 10 mg/kg within week 2. Pegylated IFN alfa2b is administered weekly at a dose of 1,5/kg/week. Patients are followed twice monthly in the first month and at least monthly thereafter (more frequently whenever is required).

Biochemical and virological assessment is recorded at week 4, 12, 24, 48. Surveillance is performed for any collateral effects and dose adjustment or growth factor need.

Ribavirin reduction is required when hemoglobin level is below 10 g/dL though EPO use.

IFN weekly administration should be reduced when neutrophiles count is < 750 in spite of G-CSF administration.

IFN interruption is required when neutrophiles are < 500 or platelets are < 35000.

End-points of the study:

* Rapid Virological Response ( week 4)
* Early Virological Response (week 12)
* Complete Early Virological Response (week 12)
* End of treatment Virological Response (week 48)
* End of treatment Biochemical Response (week 48)
* Sustained Virological Response (Six months after the end of therapy)

Collateral effects, dose adjustment and use of growth factors are recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Liver transplantation from > 6 months
2. Positive HCV-RNA viremia
3. Elevated transaminase levels (greater than 1,2 normal values) in at least two consecutive determinations during the last month
4. Histology pattern showing hepatitis C recurrence

Exclusion Criteria:

1. Multiple organ transplantation
2. Histology showing evidence of hepatic allograft rejection > 3/9 RAI score
3. Concomitant active biliary disease
4. Concomitant HBV infection
5. Normal transaminases levels
6. Less than 1500 neutrophiles in more than one blood test
7. Less than 50000 platelets in more than one blood test
8. Hemoglobin < 9 g/ dL
9. Creatinine clearance < 35 ml/min
10. Positive antibodies > 1:80
11. Auto-immune thyroid pathology
12. Severe psychiatric disease
13. Diagnosis of ischemic cardiopathy in the last 12 months
14. Active alcohol abuse
15. Low compliance to other medical treatments

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
HCV-RNA level, Transaminases level | 4°,12°,24°,36°48° week and six months after therapy conclusion

SECONDARY OUTCOMES:
liver biopsy and Transient elastography at baseline and after six month since therapy conclusion | 0°, 72° week

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Rome, Italy

REFERENCES:
- [Background] Gordon FD, Kwo P, Vargas HE. Treatment of hepatitis C in liver transplant recipients. Liver Transpl. 2009 Feb;15(2):126-35. doi: 10.1002/lt.21694. PMID 19177439
- [Background] Furusyo N, Kubo N, Toyoda K, Takeoka H, Nabeshima S, Murata M, Nakamuta M, Hayashi J. Helper T cell cytokine response to ribavirin priming before combined treatment with interferon alpha and ribavirin for patients with chronic hepatitis C. Antiviral Res. 2005 Jul;67(1):46-54. doi: 10.1016/j.antiviral.2005.04.001. PMID 15913800
- [Background] Feld JJ, Nanda S, Huang Y, Chen W, Cam M, Pusek SN, Schweigler LM, Theodore D, Zacks SL, Liang TJ, Fried MW. Hepatic gene expression during treatment with peginterferon and ribavirin: Identifying molecular pathways for treatment response. Hepatology. 2007 Nov;46(5):1548-63. doi: 10.1002/hep.21853. PMID 17929300
- [Background] Ogawa K, Hige S, Nakanishi M, Yamamoto Y, Chuma M, Nagasaka A, Asaka M. Immunological and mutagenic actions of ribavirin monotherapy preceding combination therapy with interferon for patients with chronic hepatitis C. Antivir Ther. 2009;14(4):513-22. PMID 19578236
- [Background] Tox U, Schulte S, Heindl B, Goeser T, Drebber U, Stelzer A, Steffen HM. Ribavirin priming in patients with chronic hepatitis C and normal ALT: a pilot study. Hepatogastroenterology. 2008 Sep-Oct;55(86-87):1666-70. PMID 19102366
- [Background] Cuevas JM, Gonzalez-Candelas F, Moya A, Sanjuan R. Effect of ribavirin on the mutation rate and spectrum of hepatitis C virus in vivo. J Virol. 2009 Jun;83(11):5760-4. doi: 10.1128/JVI.00201-09. Epub 2009 Mar 25. PMID 19321623
- [Background] Dixit NM, Perelson AS. The metabolism, pharmacokinetics and mechanisms of antiviral activity of ribavirin against hepatitis C virus. Cell Mol Life Sci. 2006 Apr;63(7-8):832-42. doi: 10.1007/s00018-005-5455-y. PMID 16501888
- [Background] Berenguer M. Systematic review of the treatment of established recurrent hepatitis C with pegylated interferon in combination with ribavirin. J Hepatol. 2008 Aug;49(2):274-87. doi: 10.1016/j.jhep.2008.05.002. Epub 2008 May 22. PMID 18571272
- [Background] Berenguer M, Prieto M, Rayon JM, Mora J, Pastor M, Ortiz V, Carrasco D, San Juan F, Burgueno MD, Mir J, Berenguer J. Natural history of clinically compensated hepatitis C virus-related graft cirrhosis after liver transplantation. Hepatology. 2000 Oct;32(4 Pt 1):852-8. doi: 10.1053/jhep.2000.17924. PMID 11003634
- [Background] Berenguer M, Lopez-Labrador FX, Wright TL. Hepatitis C and liver transplantation. J Hepatol. 2001 Nov;35(5):666-78. doi: 10.1016/s0168-8278(01)00179-9. No abstract available. PMID 11690716